CLINICAL TRIAL: NCT01628848
Title: A Placebo-controlled Dose-finding Study for SPM 962 in Advanced Parkinson's Disease Patients With Concomitant Treatment of L-dopa
Brief Title: A Dose-finding Study for SPM 962 in Advanced Parkinson's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 243-05-001; JapicCTI-060287 (Other: JAPIC)
Record Dates: First submitted 2012-06-24; First posted 2012-06-27 (Estimated); Results first posted 2014-03-19 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-02

CONDITIONS: Parkinson's Disease
Keywords: SPM 962; rotigotine; Parkinson's disease; concomitant use of L-dopa
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPM 962 (Experimental): SPM 962 transdermal patch
  Interventions: Drug: SPM 962
- Placebo (Placebo Comparator): Placebo transdermal patch
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPM 962 — SPM 962 transdermal patch once a daily up to 36.0 mg/day
  Arms: SPM 962
Drug: Placebo — Placebo transdermal patch
  Arms: Placebo

SUMMARY:
The primary objective of this study is to investigate efficacy and safety of SPM 962 in advanced Parkinson's Disease (PD) patients in a multi-center, placebo-controlled study following once-daily multiple transdermal doses of SPM 962 within a range of 4.5 to 36.0 mg (12 weeks of dose titration/maintenance period). Recommended maintenance dose range is also to be investigated with distribution of the maintenance dose and accumulated response rate of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Subject diagnosed as having Parkinson's disease in accordance with "Diagnostic Criteria established by the Research Committee of MHLW-specified Intractable Neurodegenerative Diseases (1995)".
* Subject is 30 and more and less than 80 years of age at the time of informed consent.
* Hoehn & Yahr stage 2-4 (on time).
* Total UPDRS Part 3 score is over 10 at screening test (on time).
* Subject is on a stable dose of L-dopa with no change in daily dose or dosing regimen for at least 28 days prior to the initial treatment of SPM 962.
* Subject has any of the following problematic symptoms; 1) Wearing off phenomenon 2) On and off phenomenon 3) Delayed-on and/or No-on phenomenon 4) Not well controlled with L-dopa due to adverse effect 5) Weakening of L-dopa efficacy.

Exclusion Criteria:

* Subject has previously participated in a trial with SPM 962.
* Subject is on other dopamine agonist treatment within 28 days prior to the initial treatment.
* Subject has psychiatric symptoms, e.g. confusion, hallucination, delusion, excitation, delirium, abnormal behavior at screening test or baseline.
* Subject has orthostatic hypotension.
* Subject has a history of epilepsy, convulsion and other.
* Subject has a complication of serious cardiac disorder or has the history.
* Subject has arrhythmia and treated with class 1a antiarrhythmic drugs (e.g. quinidine, procainamide etc.) or class 3 antiarrhythmic drugs (e.g. amiodarone, sotalol etc.).
* At screening and baseline, subject develops serious ECG abnormality. Subjects has QTc-interval >450 msec twice at screening. Subject has a the average QTc-interval from two ECGs >450 msec in males and >470 msec in females at baseline.
* Subject has congenital long QT syndrome.
* Subject has hypokalaemia.
* Subject has a total bilirubin >= 3.0 mg/dL or AST(GOT) or ALT(GPT) greater than 2.5 times of the upper limit of the reference range (or >= 100 IU/L) at screening test.
* Subject has BUN >= 25 mg/dL or serum creatinine >= 2.0 mg/dl at screening test.
* Subject has a history of allergic reaction to topical agents such as transdermal patch.
* Subject is pregnant or nursing or woman who plans pregnancy during the trial.
* Subject is receiving therapy with prohibited drug specified in the study protocol.
* Subject has a history of pallidotomy, thalamotomy, deep brain stimulation or fetal tissue transplant.
* Subject has dementia.
* Subject is unable to give consent.
* Subject is participating in another trial of an investigational drug or done so within 24 weeks prior to the initial treatment.
* Investigator judges that subject is inappropriate as a study subject with other reasons.

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2006-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyoji Imaoka, Mr, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (7):
- Japan (7):
  - Chubu Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SPM 962 | Placebo
Started | 87 | 87
Completed | 75 | 73
Not Completed | 12 | 14
Not completed — Adverse Event | 9 | 7
Not completed — Lack of Efficacy | 0 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Physician Decision | 3 | 1

BASELINE CHARACTERISTICS:
Population: Excluded 1 sebject of each arm by vaiolation of protocol
Groups:
- Total: Total of all reporting groups
Arm/Group | SPM 962 | Placebo | Total
Number analyzed (Participants) | 86 | 86 | 172
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 26 | 50
  >=65 years | 62 | 60 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (6.8) | 66.8 (8.3) | 66.9 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 42 | 94
  Male | 34 | 44 | 78
Region of Enrollment [Number; unit: participants]
  Japan | 87 | 87 | 174

OUTCOME MEASURES:

1. Primary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Part 3 Sum Score
Description: Mean change (LOCF) from baseline in UPDRS Part 3 sum score at 12 weeks after dosing.
  UPDRS is a scale for monitoring Parkinson's Disease-related disability and impairment. The UPDRS consists of the following four sub-scales. Part 1: Mentation, Part 2: Activities of Daily Living, Part 3: Motor, Part 4: Complications. Part 3 assesses 14 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: baseline, 12 weeks after dosing
Population: Full analysis set (FAS), last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962 | Placebo
Number analyzed (Participants) | 86 | 86
Scores on a scale | -10.1 (9.0) | -4.4 (7.4)

2. Secondary Outcome: UPDRS Part 2 Sum Score (Average Score of on State and Off State)
Description: Mean change (LOCF) from baseline in UPDRS Part 2 sum score (average scores of on state and off state) at 12 weeks after dosing.
  Mean change (LOCF) from baseline in UPDRS Part 2 sum score (average score of on state and off state) at 12 weeks after dosing.
  UPDRS sub-scale Part 2 assesses 13 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: baseline, 12 weeks after dosing
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962 | Placebo
Number analyzed (Participants) | 86 | 86
Scores on a scale | -3.8 (3.6) | -1.6 (2.6)

3. Secondary Outcome: Off Time
Description: Mean change (LOCF) from baseline in off time at 12 weeks after dosing.
Time Frame: baseline, 12 weeks after dosing
Population: FAS subjects with measurable off time data at baseline, LOCF
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | SPM 962 | Placebo
Number analyzed (Participants) | 54 | 56
Hours | -2.1 (3.1) | -0.7 (2.8)

4. Secondary Outcome: Effective Rate in UPDRS Part 3 Sum Score
Description: Effective rate (percentage of subjects with 20% or 30% decrease) (LOCF) in UPDRS Part 3 sum score at 12 weeks after dosing.
Time Frame: Baseline, 12 weeks after dosing
Population: FAS, LOCF
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SPM 962 | Placebo
Number analyzed (Participants) | 86 | 86
Percentage of participants
  Subjects with ≥20% decrease | 73.3 [63.9 to 82.6] | 43.0 [32.6 to 53.5]
  Subjects with ≥30% decrease | 64.0 [53.8 to 74.1] | 29.1 [19.5 to 38.7]

5. Secondary Outcome: UPDRS Part 1 Sum Score
Description: Mean change (LOCF) from baseline in UPDRS Part 1 sum score at 12 weeks after dosing.
  UPDRS sub-scale Part 1 assesses 4 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, 12 weeks after dosing
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962 | Placebo
Number analyzed (Participants) | 86 | 86
Scores on a scale | -0.15 (1.34) | -0.12 (0.79)

6. Secondary Outcome: Effective Rate in Off Time
Description: Effective rate (percentage of subjects with 20% or 30% decrease) (LOCF) in off time at 12 weeks after dosing.
Time Frame: Baseline, 12 weeks after dosing.
Population: FAS subjects with measurable off time data at baseline, LOCF
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SPM 962 | Placebo
Number analyzed (Participants) | 54 | 56
Percentage of participants
  Subjects with ≥20% decrease | 63.0 [50.1 to 75.8] | 46.4 [33.4 to 59.5]
  Subjects with ≥30% decrease | 51.9 [38.5 to 65.2] | 37.5 [24.8 to 50.2]

7. Secondary Outcome: UPDRS Part 2 Sum Score (on State)
Description: Mean change (LOCF) from baseline in UPDRS Part 2 sum score (on state) at 12 weeks after dosing.
  UPDRS sub-scale Part 2 assesses 13 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, 12 weeks after dosing
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962 | Placebo
Number analyzed (Participants) | 86 | 86
Scores on a scale | -3.0 (3.7) | -1.2 (2.6)

8. Secondary Outcome: UPDRS Part 2 Sum Score (Off State)
Description: Mean change (LOCF) from baseline in UPDRS Part 2 sum score (off state) at 12 weeks after dosing.
  UPDRS sub-scale Part 2 assesses 13 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, 12 weeks after dosing
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962 | Placebo
Number analyzed (Participants) | 55 | 59
Scores on a scale | -4.6 (4.5) | -1.9 (3.6)

9. Secondary Outcome: UPDRS Part 4 Sum Score
Description: Mean change (LOCF) from baseline in UPDRS Part 4 sum score at 12 weeks after dosing.
  UPDRS sub-scale Part 4 assesses 11 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, 12 weeks after dosing
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962 | Placebo
Number analyzed (Participants) | 86 | 85
Scores on a scale | -0.40 (1.73) | -0.22 (1.21)

10. Secondary Outcome: Total of UPDRS Part 2 Sum Score (Average Score of on State and Off State) and UPDRS Part 3 Sum Score
Description: Mean change (LOCF) from baseline in total of UPDRS Part 2 sum score (average score of on state and off state), and UPDRS Part 3 sum score at 12 weeks after dosing.
  UPDRS sub-scale Part 2 assesses 13 items and Part 3 assesses 14 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, 12 weeks after dosing
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962 | Placebo
Number analyzed (Participants) | 86 | 86
Scores on a scale | -14.0 (11.4) | -6.0 (9.3)

11. Secondary Outcome: Total of UPDRS Part 1 Sum Score, UPDRS Part 2 Sum Score (Average Score of on State and Off State), UPDRS Part 3 Sum Score, and UPDRS Part 4 Sum Score.
Description: Mean change (LOCF) from baseline in total of UPDRS Part 1 sum score, UPDRS Part 2 sum score (average score of on state and off state), UPDRS Part 3 sum score, and UPDRS Part 4 sum score at 12 weeks after dosing.
  UPDRS sub-scale Part 1, 2, 3, and 4 assess 4, 13, 14, and 11 items respectively. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, 12 weeks after dosing
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962 | Placebo
Number analyzed (Participants) | 86 | 86
Scores on a scale | -14.6 (11.9) | -6.4 (10.1)

12. Secondary Outcome: The Modified Hoehn & Yahr Severity of Illness
Description: Mean change (LOCF) from baseline in the Modified Hoehn & Yahr Severity of Illness at 12 weeks after dosing.
  The Modified Hoehn & Yahr criteria are measured on the following 8-point scale for staging: 0, No signs of disease; 1, Unilateral disease; 1.5, Unilateral plus axial involvement; 2, Bilateral disease without impairment of balance; 2.5, Mild bilateral disease with recovery on pull test; 3, Mild to moderate bilateral disease, some postural instability, physically independent 4, Severe disability, still able to walk or stand unassisted; and 5, Wheelchair bound or bedridden unless aided.
Time Frame: Baseline, 12 weeks after dosing
Population: FAS, LOCF
Measure: Number; unit: Percentage of participants
Arm/Group | SPM 962 | Placebo
Number analyzed (Participants) | 86 | 86
Percentage of participants
  Increased | 1.2 | 4.7
  Not changed | 61.6 | 80.0
  Decreased | 37.2 | 15.3

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | SPM 962 | Placebo
Serious Adverse Events (participants affected / at risk) | 3/87 | 3/87
Other Adverse Events (participants affected / at risk) | 80/87 | 59/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPM 962 (N=87) | Placebo (N=87)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hernia Inguinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Arthritis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Blood Creatine Phosphokinase Increased (Investigations) | 1 (1) | 0 (0)
Consciousness Loss (Nervous system disorders) | 0 (0) | 1 (1)
Neuroleptic Malignant (Nervous system disorders) | 1 (1) | 0 (0)
Delusion (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination, Auditory (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPM 962 (N=87) | Placebo (N=87)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 17 (17) | 5 (8)
Constipation (Gastrointestinal disorders) | 9 (9) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (10) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 4 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 1 (1)
Application Site Reaction (General disorders) | 44 (46) | 16 (21)
Application Site Erythema (General disorders) | 8 (14) | 4 (5)
Application Site Pruritus (General disorders) | 5 (5) | 4 (4)
Feeling Abnormal (General disorders) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 18 (20) | 13 (19)
Cystitis (Infections and infestations) | 2 (2) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 7 (7)
Contusion (Injury, poisoning and procedural complications) | 5 (5) | 3 (4)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Blood Creatine Phosphokinase Increased (Investigations) | 6 (6) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 4 (6) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Dyskinesia (Nervous system disorders) | 12 (13) | 7 (7)
Dizziness (Nervous system disorders) | 7 (8) | 2 (2)
Dizziness Postural (Nervous system disorders) | 7 (7) | 1 (2)
Headache (Nervous system disorders) | 5 (5) | 2 (2)
Somnolence (Psychiatric disorders) | 12 (12) | 1 (1)
Hallucination Visual (Psychiatric disorders) | 8 (10) | 2 (2)
Hallucination (Psychiatric disorders) | 3 (3) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3) | 3 (3)
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No